CLINICAL TRIAL: NCT00129441
Title: Treatment of Cognitive Disability in Schizophrenia With a GABA-A Alpha2/3 Receptor Agonist
Brief Title: Gamma-Amino Butyric Acid (GABA)-A Alpha2/3 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0502027
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Merck L-830982 (Experimental)
  Interventions: Drug: Merck L-830982
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Merck L-830982 — The initial dose of L-830982 was 3.0 mg twice daily (b.i.d.) the dosage increased to 5.0 mg b.i.d. at the end of week 1 and 8.0 mg b.i.d. at the end of week 2, which was continued for the remaining 2 weeks of the trial. Medications were dispensed weekly in blister packs by the hospital pharmacy.
  Other Names: MK-0777
  Arms: Merck L-830982
Drug: Placebo — Medications were dispensed weekly in blister packs by the hospital pharmacy, using the same number of pills as those on active drug.
  Arms: Sugar pill

SUMMARY:
The purpose of this research study is to determine whether a short-term administration of an investigational study drug may provide evidence of improvement in cognitive functioning in a group of stable male subjects with schizophrenia.

DETAILED DESCRIPTION:
The goal of this study is to determine whether the short-term (4 week), double-blind administration of Merck L-830982 provides evidence of improvement in cognitive functioning in stable male subjects with schizophrenia. This initial, small sample size study (n=9 on L-830982 and n=6 on placebo) is restricted to males in order to reduce the variance that might be attributable to the well-documented sex differences in the clinical features of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Between the ages of 18 and 50
* Meet diagnostic criteria for schizophrenia or schizoaffective disorder
* Are clinically stable for a minimum of 3 months on current dose of medication
* Are unemployed (i.e., work less than 20 hours per week at competitive employment)

Exclusion Criteria:

* Psychoactive substance dependence within the past 6 months or substance abuse within the past month
* History of head trauma or other neurological disorder
* Medical illness or medications, such as benzodiazepine treatment or HIV medications, that may be affected by study participation (the study doctor will discuss this with potential subjects)
* Mental retardation
* Seizure disorder
* History of a heart attack, arrhythmia, or other heart disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Lewis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Lewis DA, Hashimoto T, Volk DW. Cortical inhibitory neurons and schizophrenia. Nat Rev Neurosci. 2005 Apr;6(4):312-24. doi: 10.1038/nrn1648. PMID 15803162
- [Background] Lewis DA, Volk DW, Hashimoto T. Selective alterations in prefrontal cortical GABA neurotransmission in schizophrenia: a novel target for the treatment of working memory dysfunction. Psychopharmacology (Berl). 2004 Jun;174(1):143-50. doi: 10.1007/s00213-003-1673-x. Epub 2003 Dec 9. PMID 15205885
- [Result] Lewis DA, Cho RY, Carter CS, Eklund K, Forster S, Kelly MA, Montrose D. Subunit-selective modulation of GABA type A receptor neurotransmission and cognition in schizophrenia. Am J Psychiatry. 2008 Dec;165(12):1585-93. doi: 10.1176/appi.ajp.2008.08030395. Epub 2008 Oct 15. PMID 18923067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through referrals from clinicians in the outpatient clinical services at Western Psychiatric Institute & Clinic and through a Psychosis Registry. 29 males signed consent and 16 were eligible-one subject did not complete the study and is not included in any summary statistics. Recruitment period: 4/05 through 1/07.
Pre-assignment Details: To ensure eligibility before randomization, the following were administered: a urine drug screen; diagnostic, medical history and adverse events ratings; Repeatable Battery for the Assessment of Neuropsychological Status (RBANS); electrocardiogram; blood tests (for kidney and liver function); and a complete eye exam, including a slit-lamp exam.
Groups:
- L-830982: The initial dose of L-830982 was 3.0 mg twice daily (b.i.d.) the dosage increased to 5.0 mg b.i.d. at the end of week 1 and 8.0 mg b.i.d. at the end of week 2, which was continued for the remaining 2 weeks of the trial. Medications were dispensed weekly in blister packs by the hospital pharmacy.
Period: Overall Study
Arm/Group | L-830982 | Placebo
Started | 9 | 6
Baseline, Visit 1 | 9 (Baseline # only includes those who completed 4-week trial (one L-830982 subject did not complete).) | 6
Week 1, Visit 2 | 9 | 6
Week 2, Visit 3 | 9 | 6
Week 3, Visit 4 | 9 | 6
Week 4, Visit 5 | 9 | 6
Week 5, Visit 6 | 9 | 6
Week 26, Visit 7 | 9 | 6
Year 1, Visit 8 | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-830982 | Placebo | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.6) | 35.7 (6.8) | 37.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: Participants]
  United States | 9 | 6 | 15
N-back Task Reaction Time [Mean (Standard Deviation); unit: msec] — The N-back task is a sequential-letter memory task for which working memory load is varied, as the respondent must indicate when the current stimulus matches the one from 'n' steps earlier in the sequence. Those with schizophrenia exhibit substantially impaired performance and decreased functional activation of the dorsolateral prefrontal cortex (DLPFC) relative to matched comparison subjects for the 2-back load condition. 2-back condition was used as the dependent measure, as it provides the best index of performance and DLPFC disturbances in subjects with schizophrenia.
  msec | 874 (238) | 669 (158) | 801 (230)
N-back Task Error Rate [Mean (Standard Deviation); unit: proportion of errors] — The N-back task is a sequential-letter memory task for which working memory load is varied, as the respondent must indicate when the current stimulus matches the one from 'n' steps earlier in the sequence. Those with schizophrenia exhibit substantially impaired performance and decreased functional activation of the dorsolateral prefrontal cortex (DLPFC) relative to matched comparison subjects for the 2-back load condition. 2-back condition was used as the dependent measure, as it provides the best index of performance and DLPFC disturbances in subjects with schizophrenia.
  proportion of errors | 0.247 (0.102) | 0.250 (0.028) | 0.248 (0.081)
AX Continuous Performance Test Task d-prime [Mean (Standard Deviation); unit: d-prime] — For the AX Continuous Performance Test (AXCPT), subjects are required to maintain an attentional set across a delay interval in order to overcome a prepotent response tendency (target responses are required when an X is presented but only in the context of a preceding A; non-target conditions are AY, BX and BY). The dependent measure was d-prime at the long delay (calculated as AX hits minus BX false alarms, which is particularly sensitive to context processing impairments in individuals with schizophrenia.
  d-prime | 0.9 (0.7) | 0.7 (0.9) | 0.8 (0.7)
Preparing to Overcome Prepotency (POP) Task - Reaction Time [Mean (Standard Deviation); unit: msec] — The POP task is a cued stimulus-response reversal paradigm that, similar to the AX Continuous Performance Test, requires increases in cognitive control through the maintenance and use of context information to overcome prepotent response tendencies.
  msec | 66 (48) | 36 (61) | 54 (53)
Preparing to Overcome Prepotency (POP) Task - Error Rate [Mean (Standard Deviation); unit: proportion of errors] — The POP task is a cued stimulus-response reversal paradigm that, similar to the AX Continuous Performance Test, requires increases in cognitive control through the maintenance and use of context information to overcome prepotent response tendencies.
  proportion of errors | 0.034 (0.050) | 0.064 (0.068) | 0.046 (0.058)
Brief Psychiatric Rating Scale (BPRS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Brief Psychiatric Rating Scale-anchored (BPRS; Overall and Gorham, 1962; Woerner, Mannuzza, Kane, 1988) is an 18-item scale that is among the most widely used measure of psychopathology. Scores range from 1-7, with higher scores reflecting greater pathology. A total score is derived from the sum of all 18 items (possible scores range from 18-126). It relies on clinical judgment in the assessment of key areas of psychopathology (depression, anxiety, psychosis).
  Scores on a scale | 24.3 (2.6) | 34.2 (7.1) | 28.3 (6.9)
Repeatable Battery for the Assessment of Neuropsychological Status: RBANS Total Score [Mean (Standard Deviation); unit: Standard Score] — Five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score. The Total Score is expressed as a standardized score normalized to a population mean of 100, with a standard deviation of 15 (possible scores 40-135). Higher scores reflect better performance. All subjects received the "A" form at baseline and the wk-4 visit and the "B" form at the wk-2 visit (the A/B forms are equivalent alternate forms, which allow for retesting patients without the confound of practice effects).
  Standard Score | 71.8 (10.6) | 63.5 (7.1) | 68.5 (10.0)
Repeatable Battery for the Assessment of Neuropsychological Status: RBANS Delayed Memory Subindex [Mean (Standard Deviation); unit: Standard Score] — The Delayed Memory Index consists of verbal and nonverbal recall tasks (words, drawings) that the subject views early in the evaluation and without warning, is asked to recall ~1/2 hr later. Scores are expressed as standardized scores normalized to a population mean of 100, with a standard deviation of 15 (possible scores between 40-135). Higher scores reflect better performance. Subjects received the "A" form at baseline and wk-4 visit and the "B" form at the wk-2 visit (A/B forms are equivalent alternate forms, which allow for retesting patients without the confound of practice effects).
  Standard Score | 76.8 (15.5) | 60.8 (16.1) | 70.4 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: N-back Task - Reaction Time
Description: The N-back task is a sequential-letter memory task for which working memory load is varied, as the respondent must indicate when the current stimulus matches the one from 'n' steps earlier in the sequence. The dependent measure for the N-back task was performance in the 2-back condition, which provides the best index of performance and dorsolateral prefrontal cortex disturbances in subjects with schizophrenia.
Time Frame: Week 4
Population: Analyses included only those participants who completed the 4-week trial. One participant refused N-back at week-4, so 9 L-830982 and 5 placebo were analyzed.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 5
msec | 786 (231) | 684 (101)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p = 0.16, ANOVA

2. Primary Outcome: N-back Task - Error Rate
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of errors
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 5
proportion of errors | 0.239 (0.062) | 0.297 (0.075)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p = 0.162, ANOVA

3. Primary Outcome: AX Continuous Performance Test Task D-prime
Description: For the AX Continuous Performance Test, subjects are required to maintain an attentional set across a delay interval in order to overcome a prepotent response tendency (target responses are required when an X is presented but only in the context of a preceding A; non-target conditions are AY, BX and BY). The dependent measure was d-prime at the long delay (calculated as AX hits minus BX false alarms, which is particularly sensitive to context processing impairments in individuals with schizophrenia.
Time Frame: Week 4
Population: Four subjects did not complete a sufficient number of trials for the AXCPT task at both testing periods, therefore 7 L-830982 and 4 placebo subjects data were analyzed.
Measure: Mean (Standard Deviation); unit: d-prime
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 7 | 4
d-prime | 1.9 (0.9) | 0.7 (0.9)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p = 0.12, ANOVA

4. Primary Outcome: Preparing to Overcome Prepotency (POP) Task - Reaction Time
Description: The POP task is a cued stimulus-response reversal paradigm that, similar to the AX Continuous Performance Test, requires increases in cognitive control through the maintenance and use of context information to overcome prepotent response tendencies.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 6
msec | 57 (66) | 66 (55)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p = 0.05, ANOVA

5. Primary Outcome: Preparing to Overcome Prepotency Task - Error Rate
Description: as for outcome 4
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: proportion of errors
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 6
proportion of errors | 0.042 (0.042) | 0.031 (0.074)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p = 0.249, ANOVA

6. Secondary Outcome: Brief Psychiatric Rating Scale Total Score
Description: The Brief Psychiatric Rating Scale-anchored (BPRS; Overall and Gorham, 1962; Woerner, Mannuzza, Kane, 1988) is an 18-item scale that is among the most widely used measure of psychopathology. Scores range from 1-7, with higher scores reflecting greater pathology. A total score is derived from the sum of all 18 items (possible scores range from 18-126). It relies on clinical judgment in the assessment of key areas of psychopathology (depression, anxiety, psychosis).
Time Frame: Week 4
Population: One subject dropped out prior to completing study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 6
Scores on a scale | 26.3 (5.3) | 27.0 (3.0)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; At week 4, mean BPRS total scores were nearly the same for the placebo group and L-830982 group as a result of a significant reduction in positive symptoms reported for the placebo group (F=9.12, df=1,13, p=0.01). For the L-830982-treated group, neither total BPRS scores nor any of the factor scores changed over the course of the trial; Test type: Superiority or Other; p = 0.01, ANOVA

7. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Score
Description: Five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score. The Total Score is expressed as a standardized score normalized to a population mean of 100, with a standard deviation of 15 (possible scores 40-135). Higher scores reflect better performance. All subjects received the "A" form at baseline and the wk-4 visit and the "B" form at the wk-2 visit (the A/B forms are equivalent alternate forms, which allow for retesting patients without the confound of practice effects).
Time Frame: Week 4
Population: One subject dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: Standard Score
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 6
Standard Score | 76.7 (13.5) | 70.8 (12.4)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status - Delayed Memory Subindex
Description: The Delayed Memory Index consists of verbal and nonverbal recall tasks (words, drawings) that the subject views early in the evaluation and without warning, is asked to recall ~1/2 hr later. Scores are expressed as standardized scores normalized to a population mean of 100, with a standard deviation of 15 (possible scores between 40-135). Higher scores reflect better performance. Subjects received the "A" form at baseline and wk-4 visit and the "B" form at the wk-2 visit (A/B forms are equivalent alternate forms, which allow for retesting patients without the confound of practice effects).
Time Frame: Week 4
Population: One subject dropped out before completing the study.
Measure: Mean (Standard Deviation); unit: Standard Score
Arm/Group | L-830982 | Placebo
Number analyzed (Participants) | 9 | 6
Standard Score | 85.3 (15.7) | 63.8 (17.6)
Statistical Analysis 1: Comparison: L-830982 vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at all timepoints during the 5-week clinical trial. Eye exams were conducted at 6-month and 1-year follow-ups.
Arm/Group | L-830982 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-830982 (N=10) | Placebo (N=6)
Dizziness (General disorders) | 2 (2) | 0 (0)
Somnolence (General disorders) | 2 (2) | 0 (0)
Appetite increase (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size; RBANS may lack appropriate sensitivity for short-term study; between-group differences in baseline clinical symptoms & neuropsychological function; excluding those with more modest cognitive impairments (RBANS standard score >90).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No